CLINICAL TRIAL: NCT05903846
Title: The Effect of Oketani Massage on Breastfeeding Success and Breast Engorgement in Mothers Delivering by Cesarean Section: A Randomized Controlled Study
Brief Title: The Effect of Oketani Massage on Breastfeeding Success and Breast Engorgement in Mothers Delivering by Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Emine Serap ÇAĞAN, assistant professor, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AgriIbrahimCecenU
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2023-06

CONDITIONS: Breastfeeding; Engorgement of Breast Associated With Childbirth, Postpartum
Keywords: breastfeeding; Engorgement; Oketani massage
MeSH Terms: conditions — Breast Feeding; Hyperemia

STUDY DESIGN:
Intervention Model Description: Oketani massage,The part between the breast and the base of the lower pectoral muscle is called the "oketani". It is a manual massage technique developed to encourage breastfeeding in breastfeeding problems such as insufficient milk production and mastitis. It is a massage that stimulates the breast, relaxes it and is painless. There are 8 different stages in massage. Each set lasts 1 minute, the massage continues for 15-20 minutes.
Who Masked: Outcomes Assessor
Masking Description: Massage was applied to the Oketani massage group by a midwife working in the clinicThe outcome assessor does not know who the groups are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oketani massage group (Experimental): According to the Ministry of Health, the follow-up period for mothers after cesarean section in Turkey is 48 hours. After the mothers in the massage group were taken to the service, oketani massage was applied three times a day for an average of 15-20 minutes, starting before breastfeeding. Massage was applied to the Oketani massage group by a midwife working in the clinic. Before the mothers were discharged, the breast fullness and breastfeeding status of the mothers were evaluated using the breast engorgement assessment scale and the LATCH breastfeeding diagnostic scale.
  Interventions: Other: Oketani massage
- Control group (No Intervention): No intervention was made in the control group and routine follow-up of mothers and babies will be performed after cesarean section. No intervention was made regarding the breastfeeding process of the mothers, other than the breastfeeding counseling given by the breastfeeding consultant according to the hospital protocol. Before the mothers were discharged, the breast fullness and breastfeeding status of the mothers were evaluated using the breast fengorgement assessment scale and the LATCH breastfeeding diagnostic scale.

INTERVENTIONS:
Other: Oketani massage — The part between the breast and the base of the lower pectoral muscle is called the "oketani". It is a manual massage technique developed to encourage breastfeeding in breastfeeding problems such as insufficient milk production and mastitis. It is a massage that stimulates the breast, relaxes it and is painless.
  Arms: Oketani massage group

SUMMARY:
The aim of this study was to examine the effect of octani massage on breastfeeding success and breast engorgement in mothers who gave birth by cesarean section. The research was carried out in the gynecology service of Ağrı Training and Research Hospital between November 2022 and April 2023. The universe of the study consisted of mothers who were hospitalized in the gynecology service of Ağrı Training and Research Hospital between November 2022 and April 2023 and gave birth by cesarean section. The Open Epi calculation tool was used to determine the sample of the study. The sample calculation was made on the average score differences in the Open Epi info program. Accordingly, it was planned to include 106 mothers, 53 of whom were in the control group and 53 in the massage group. Considering the sample loss to be experienced during data collection, a total of 116 mothers, 58 in the control group and 58 in the massage group, were included in the study. Randomization of the groups participating in the study was made as simple randomization using the www.random.org site. Introductory Characteristics Questionnaire, oketany massage follow-up form, breast engorgement assessment scale and LATCH breastfeeding diagnostic measurement tool were used to collect the research data.

DETAILED DESCRIPTION:
The research was carried out in two groups, namely the octopus massage group and the control group.

Oketani Massage Group: According to the Ministry of Health, the follow-up period for mothers after cesarean section in Turkey is 48 hours. After the mothers in the massage group were taken to the service, oketani massage was applied three times a day for an average of 15-20 minutes, starting before breastfeeding. Massage was applied to the Oketani massage group by a midwife working in the clinic. Before the mothers were discharged, the breast engorgement and breastfeeding status of the mothers were evaluated using the breast fullness assessment scale and the LATCH breastfeeding diagnostic scale. Control Group: No intervention was made in the control group and routine follow-up of mothers and babies will be performed after cesarean section. No intervention was made regarding the breastfeeding process of the mothers, other than the breastfeeding counseling given by the breastfeeding consultant according to the hospital protocol. Before the mothers were discharged, the breast engorgement a and breastfeeding status of the mothers were evaluated using the breast fullness assessment scale and the LATCH breastfeeding diagnostic scale.

ELIGIBILITY:
Inclusion criteria for the study:

* Delivery by cesarean section
* Single and live birth,
* 38-40 Giving birth between weeks
* Not having a mental or physical disability that prevents breastfeeding,
* The baby does not need neonatal intensive care
* The baby does not have a condition that prevents breastfeeding
* Sharing the same room with the baby
* Agreeing to participate in the research

Exclusion criteria from the study:

* Refusal to participate in the study
* Giving birth normally
* Giving birth prematurely
* Having a mental and physical disability that prevents breastfeeding
* Being 18 years of age or younger
* Transferring the baby to the neonatal intensive care unit
* Having a condition that prevents breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers giving birth and breastfeeding were included in the study.
Enrollment: 116 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Breast engorgement assessment scale | postpartum 48 hours from birth
  The scale is scored from 1 to 6. On the scale, "1" is evaluated as no soft change, while "6" is expressed as very hard and very sensitive. If the score from the scale is higher than 4, it means that there is breast fullness.
LATCH breastfeeding diagnostic scale | postpartum 48 hours from birth
  by observing breastfeeding; It is an assessment tool that is quick and easy to apply, created to detect problems that may occur during breastfeeding. Scoring is done between 0-2 and the maximum score that can be obtained is 10. In the non-breakpoint measurement tool, a high score indicates successful breastfeeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Agri Ibrahim Cecen University, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided